CLINICAL TRIAL: NCT02857569
Title: A Randomized Phase I/II Trial Evaluating the Safety & Efficacy of Intra-Tumoral Ipilimumab in Combination With Intra-venous Nivolumab in Patients With Metastatic Melanoma
Brief Title: A Trial Evaluating the Safety & Efficacy of Intra-Tumoral Ipilimumab in Combination With Intra-venous Nivolumab in Patients With Metastatic Melanoma
Acronym: NIVIPIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-005429-37; 2015/2334 (Other: CSET Number)
Record Dates: First submitted 2016-07-19; First posted 2016-08-05 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Stage III/IV Melanoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental IT Arm (Experimental): * ipilimumab: 0.3mg/kg IT injection every 3 weeks until complete response, eradication of all injectable sites, disease progression or toxicity, for a maximum of 4 doses (to compare back to back to IV standard of care and marketing authorization).
  * nivolumab: 1mg/kg, IV injection every 3 weeks during IT ipilimumab treatment period and 3mg/kg, IV injection every 2 weeks after IT ipilimumab treatment interruption. Treatment should be continued as long as clinical benefit is observed or until treatment is no longer tolerated by the patient for a maximum of 12 months.
  Interventions: Drug: Ipilimumab IT; Drug: Nivolumab IV
- Standard Arm (Active Comparator): * ipilimumab: 3mg/kg, IV injection every 3 weeks for a maximum of 4 doses as per standard of care and marketing authorization.
  * nivolumab: 1mg/kg, IV injection every 3 weeks during IV ipilimumab treatment period and 3mg/kg, IV injection every 2 weeks after IV ipilimumab treatment interruption. Treatment should be continued as long as clinical benefit is observed or until treatment is no longer tolerated by the patient for a maximum of 12 months.
  Interventions: Drug: Ipilimumab IV; Drug: Nivolumab IV

INTERVENTIONS:
Drug: Ipilimumab IT
  Arms: Experimental IT Arm
Drug: Ipilimumab IV
  Arms: Standard Arm
Drug: Nivolumab IV

SUMMARY:
The study aims to evaluate the 6 month-treatment tolerance defined as the immune related grade 3-4 adverse event-free survival of the combination therapy IT ipilimumab + IV nivolumab.

The IV ipilimumab + IV nivolumab (same doses than in Phase I) arm will be used as an internal control to interpret the results obtained in the IT ipilimumab arm.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women >/= 18 years of age
2. Signed and dated written informed consent prior any study related procedure
3. Histologically confirmed and clinically or radiologically progressing unresectable Stage III or Stage IV melanoma, as per AJCC staging system
4. Patients with at least two lesions:

   * At least one injectable tumor lesion (≥1cm3)
   * At least one target lesion (measurable lesion as per RECIST 1.1)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Treatment naïve subjects or patients relapsing after prior local or systemic anticancer therapy. Note that systemic anticancer therapy is permitted if it was completed at least 28 days or 5 times its half life (whichever is shorter) prior to the first study dose, and all related adverse events have either returned to baseline or stabilized.
7. Measurable disease by CT or MRI per RECIST 1.1 criteria.
8. Recent (less than 3 month) tumor tissue must be provided for patient stratification and biomarker analyses. In order to be equally randomized, a subject must be classified as PDL1 positive, PD-L1 negative, or PD-L1 indeterminate. If an insufficient amount of tumor tissue is available prior to the start of the screening phase, subjects must consent to allow the acquisition of additional tumor tissue for performance of biomarker analyses.
9. Subjects with wild-type BRAF. BRAF-mutant can be included only if they have been treated with, or developed toxicity with or refused to be treated with BRAF-and/or MEK-targeted therapy in front-line
10. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration.
11. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

    * WBC >/= 2000/μL
    * Neutrophils >/= 1500/μL
    * Platelets >/= 100 x103/μL
    * Hemoglobin >/= 9.0 g/dL
    * Serum creatinine </= 1.5 x ULN or creatinine clearance (CrCl) >/= 40 mL/min (using the Cockcroft-Gault formula):

    Female CrCl = [(140 - age in years) x weight in kg x 0.85] / (72 x serum creatinine in mg/dL) Male CrCl = [(140 - age in years) x weight in kg x 1.00] / (72 x serum creatinine in mg/dL)
    * AST and ALT ≤3.0 x upper limit of normal (ULN); if liver metastases AST and ALT ≤5.0 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
12. Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (ie, subject has not been randomized / has not been treated) after obtaining agreement from the coordinator prior to re-enrolling a subject. If re-enrolled, the subject must be re-consented.
13. Women of childbearing potential (WOCBP) must have a negative serum β-HCG pregnancy test within 7 days prior to initiation of treatment. Both sexually active females and males (and their female partners) patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 5 months after last study drug administration
14. Patients must be willing and able to comply with the visits, treatments, procedures, and laboratory tests, and other requirements that are scheduled in the protocol.
15. Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases or leptomeningeal disease are eligible if these lesions have been treated or if they are asymptomatic and there is no clinical evidence of progression within 28 days prior to first dose of study drug administration. CNS lesions should be monitored bu contrast enhanced MRI at disease assessment timepoints. Justification for allowing patient with CNS disease: whereas tumor-targeting antibodies have limited access to the central nervous system because of the blood brain barrier, immune targeted antibodies can generate a T-cell mediated anti-tumor immune response which I able to cross the blood brain barrier. Indeed, anti-CTLA-4 and anti PD-1 imAbs have shown their ability to induce tumor responses from metastatic sites all over the body, including in the brain
2. Ocular melanoma. Distant metastatic relapse of ocular melanoma outside the CNS can be discussed with the study coordinator on a case by case basis.
3. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
4. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
5. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
6. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
8. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
9. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. History of allergy to study drug components.
11. History of severe hypersensitivity reaction to any monoclonal antibody.
12. Pregnancy or breastfeeding
13. Patients presenting coagulation abnormalities and/or patients requiring concomitant treatment with therapeutic doses of anticoagulants. Prophylactic low dose of anticoagulants for thrombo-embolic events is allowed. Prophylactic anticoagulants shall be stopped during 24h prior and after deep lesion biopsies/injections. No stopping rule for biopsies/injections of skin and sub-cutaneous lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
6-months treatment-related grade 3-4 toxicity event-free survival (EFS). | Assessed every 28 days after randomization up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No